CLINICAL TRIAL: NCT01104116
Title: Utility of [18F]-FDG PET Imaging to Distinguish Malignant From Benign Intrapapillary Mucinous Neoplasms
Brief Title: Use of PET Imaging to Distinguish Malignant From Benign IPMN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment; PI left the institution
Sponsor: Columbia University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAD9508; UL1RR024156 (NIH)
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasm; Pancreatic Cancer
Keywords: Pancreatic Cancer; Intraductal Papillary Mucinous Neoplasm; Pre-cancerous pancreatic lesion; PET Scan; Pancreatic Cancer Screening
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/CT imaging (Experimental): Surgical patients will undergo [18F]-FDG PET/CT imaging
  Interventions: Radiation: [18F]-FDG PET/CT imaging

INTERVENTIONS:
Radiation: [18F]-FDG PET/CT imaging — Drug: F-18 Fluoro-2-Deoxyglucose (F-18 FDG)

SUMMARY:
Intraductal papillary mucinous neoplasm (IPMN) is a cystic pancreatic lesion that is a precursor to invasive pancreatic cancer. Differentiating whether an IPMN lesion is benign or malignant is critical, as the prognosis and management differs drastically, varying from surgery to clinical observation. However, despite physicians' attempts to characterize features concerning for malignancy, it is difficult to determine the likelihood of malignancy with conventional imaging techniques, and an accurate and non-invasive test to identify malignant IPMN is needed. Our hypothesis is that positron emission tomography (PET), a three-dimensional imaging that can identify cancer cells through their increased use of sugars, may be a superior test for differentiating between benign and malignant IPMN lesions. The investigators are planning a prospective pilot study of patients with IPMN who are undergoing surgery for their disease. These patients will undergo PET imaging, as well as computed tomography (CT), magnetic resonance imaging (MRI), and endoscopic ultrasound (EUS) as clinically indicated. Samples of tissue removed during surgery will be assessed and will serve as the gold standard for determining whether the lesion is benign or malignant. The investigators will evaluate the positive and negative predictive values of PET imaging for malignancy within IPMN lesions.

DETAILED DESCRIPTION:
Intraductal papillary mucinous neoplasm (IPMN) is a cystic pancreatic neoplasm that is a precursor to invasive pancreatic cancer. Differentiating whether an IPMN lesion is benign or malignant is critical, as the prognosis and management differs drastically, varying from surgical resection to observation. However, despite attempts to characterize features concerning for malignancy, it is difficult to determine the likelihood of malignancy with conventional imaging techniques, including CT, MRI, and EUS. An accurate, non-invasive test to identify malignant IPMN is needed.

The investigators' hypothesis is that [18F]-FDG PET may be a superior modality for differentiating between benign and malignant IPMN lesions. We are planning a prospective pilot study of ten consecutive patients with IPMN from the Columbia University Pancreas Center who are undergoing surgical resection for their disease. These patients will undergo [18F]-FDG PET imaging, as well as CT, MRI, and EUS as clinically indicated. All scans will be reviewed by two experienced nuclear medicine radiologists who will be blinded to the clinical characteristics of study patients and who will reach a consensus. Areas of focally increased [18F]-FDG intake will be identified. Side-by-side reading with CT scan will be performed to evaluate whether the increased [18F]-FDG uptake corresponds to a pancreatic lesion. Mean and maximal standardized uptake value (SUV) values, as well as differences in intensity between the region of interest and the remaining pancreas, will be calculated.Surgical pathology will be utilized as the gold standard for histological determination. Standard post-operative histological interpretation of each IPMN lesion will be recorded, including size, duct involvement (main, side, or mixed), ductal dilatation, lesion location (head, neck, body, tail), and histologic grade (adenoma, borderline, carcinoma in situ, invasive carcinoma). In addition, any associated pancreatitis or any other non-IPMN neoplastic change will also be noted.

Using PET scan results and surgical pathology information, we will evaluate the positive and negative predictive values of [18F]-FDG PET for malignancy within IPMN lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is seen in consultation for IPMN at Columbia-Presbyterian Medical Center and scheduled for surgical resection.
* Patient has radiological evidence, by CT or MRI, suspicious for IPMN, with cystic lesion involving main duct of size equal to or greater than 3 cm and/or involvement of at least a 3 cm segment of the main pancreatic duct.
* Patient has undergone EUS with aspiration of cyst fluid with sufficient fluid for CEA level.
* Patient is at least 18 years of age.
* Patient is able to provide written, informed consent.

Exclusion Criteria:

* Active pancreatitis within 30 days of recruitment.
* Uncontrolled diabetes mellitus.
* Pregnancy or breastfeeding (urine beta-HCG will be performed on all women of child-bearing age prior to enrollment in study).
* Unwillingness or inability to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya Divgi, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Data will not be analyzed. Only the demographic information on 1 enrolled subject is available.
Period: Overall Study
Arm/Group | PET/CT Imaging
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PET/CT Imaging
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Predictive Value of PET Imaging for Identifying Malignant IPMN
Description: The primary outcome will be to determine the positive and negative predictive values of [18F]-FDG PET imaging for identifying malignant IPMN lesions in patients who are to undergo surgical resection. We will determine the mean SUV that would provide optimal positive predictive value for malignant IPMN. IPMN lesions will be classified categorically as benign (adenoma or borderline ) or malignant (in situ or invasive carcinoma) and PET imaging will be classified categorically as negative or positive, with focal FDG uptake corresponding to pancreatic lesion.
Time Frame: 1 month
Population: The principal investigator has left the institution. Data will not be analyzed. Only the demographic information on 1 enrolled subject is available.
Arm/Group | PET/CT Imaging
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Lesion Characteristics to Assess Benefit of PET Scans
Description: The secondary outcome that we are interested in studying is the benefit of PET scan as compared to other imaging modalities, such as CT, MRI, and EUS. Thus, Patients will also have CT, MRI, and EUS imaging. We will look at how size, location, and branch of the IPMN lesion on PET compare to these other imaging modalities. The location, size, and pathology results of the actual surgical specimen will serve as the gold standard.
Time Frame: 1 month
Population: as for outcome 1
Arm/Group | PET/CT Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Data will not be analyzed. Only the demographic information on 1 enrolled subject is available.
Arm/Group | PET/CT Imaging
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No